CLINICAL TRIAL: NCT05981144
Title: Exploration of Clonal Hematopoiesis of Indeterminate Potential in Non-ischemic Heart Failure With Reduced Ejection Fraction
Status: Completed | Type: Observational
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Other Study IDs: 4-2021-0921
Record Dates: First submitted 2023-07-31; First posted 2023-08-08 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Heart Failure With Reduced Ejection Fraction

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Experimental: Patients with heart failure without significant stenosis of the major epicardial coronary artery and reduced left ventricular ejection fraction below 40%

SUMMARY:
Clonal hematopoiesis of indeterminate potential (CHIP) refers to a phenomenon in which blood cells with somatic mutation circulate in the peripheral blood due to abnormal proliferation and differentiation of mutant hematopoietic cells.

CHIP is considered one of the aging phenomena, and the mutant blood cells increased by CHIP cause chronic inflammation, thereby increasing the occurrence of atherosclerotic cardiovascular disease. Therefore, CHIP is known to be closely related to poor prognosis of ischemic heart failure. Meanwhile, chronic inflammation may be involved in the development of non-ischemic myocardial disease, which is one of the major causes of heart failure.

This study will identify CHIP and perform NLRP3 inflammasome assay in 100 non-ischemic heart failure patients and evaluate the relationship between CHIP and inflammation, imaging markers of heart failure, Left ventricle reverse remodeling after guideline-directed medical treatment, and prognosis of heart failure with reduced ejection fraction.

ELIGIBILITY:
Inclusion Criteria:

1. As an adult over the age of 19
2. A history of left ventricular ejection fraction less than 40% on imaging tests within 3 years (HFrEF diagnosis),
3. Have a cardiac MRI taken within 3 months of being diagnosed with HFrEF,
4. A person who was diagnosed with non-ischemic heart failure by performing coronary artery imaging (angiography, CT) at the time of diagnosis of HFrEF

Exclusion Criteria:

1. Patients with confirmed ischemic cardiomyopathy (when stenosis of 75% or more of major coronary arteries is confirmed on coronary artery imaging or ischemic cardiomyopathy findings such as transmural late gadolinium enhancement on cardiac MRI)
2. History of solid cancer diagnosis and chemotherapy (drugs, radiation)
3. History of blood cancer

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients who need ACEI for cardiovascular disease
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2021-11-23 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Left ventricular reverse remodeling | 3 months after guideline-directed medical treatment
  a second measurement of left ventricular ejection fraction > 40% and a ≥10% increase from baseline left ventricular ejection fraction of ≤ 40%

SECONDARY OUTCOMES:
Clinical outcome | 3 years after enrollment
  Heart failure hospitalization or cardiovascular death

CONTACTS AND LOCATIONS:
Overall Officials: Chan Joo Lee, Principal Investigator — Division of Cardiology, Severance Hospital, Yonsei University College of Medicine
Locations (1):
- Severance hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: Undecided